CLINICAL TRIAL: NCT00512902
Title: Pilot Study to Examine The Use of Imatinib (Gleevec) For The Treatment of Active Alveolitis in Systemic Sclerosis
Brief Title: A Study Using The Experimental Drug Called Imatinib (Gleevec) in Subjects With Systemic Sclerosis
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: University of California, Los Angeles (Other)
Collaborators: Novartis Pharmaceuticals (Industry)
Responsible Party: Principal Investigator, Daniel Furst, M.D., Carl M Pearson Professor of Rheumatology, University of California, Los Angeles
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CST1571EUS210
Record Dates: First submitted 2007-08-06; First posted 2007-08-08 (Estimated); Results first posted 2014-10-27 (Estimated); Last update posted 2014-10-27 (Estimated); Status verified 2014-10

CONDITIONS: Alveolitis; Systemic Sclerosis
Keywords: active alveolitis in systemic sclerosis
MeSH Terms: conditions — Scleroderma, Systemic | interventions — Imatinib Mesylate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Group 1 (Experimental): SSc patients receiving Imatinib (Gleevec, up to 600 mg) QD PO for up to 1 year.
  Interventions: Drug: Imatinib

INTERVENTIONS:
Drug: Imatinib — All subjects will receive gleevec. Subjects will have a clinic visit every 2 weeks for the first 20 weeks and then they will have one every 4 weeks for the remainder of the study. Gleevec will be taken by mouth everyday. It will be increased to a maximum of 600 mg every day. It will be increased 100 mg at each visit for the first 12 weeks. Your participation may last up to 1 year and participants will have approximately 18 clinic visits.
  Other Names: Gleevec
Drug: Imatinib — Up to 600 mg QD PO for up to 1 year.
  Other Names: Gleevec

SUMMARY:
The purpose of this study is to assess the safety and tolerability of imatinib (gleevec) in subjects who have systemic sclerosis. Imatinib has been approved by the FDA for the treatment of newly diagnosed adult patients with CML (newly diagnosed adult patients and for the treatment of patients with an accelerated phase. Imatinib is also approved for the treatment of patients with a certain type of gastrointestinal cancer (called stromal tumors) but it has not been approved to treat systemic sclerosis. Imatinib works by interfering with an enzyme called tyrosine phosphatase resulting in suppression of the immune system. It als interferes with a protein called platelet derived growth factor receptor (PDGFr) that has been linked to increased fibrosis.

DETAILED DESCRIPTION:
Systemic sclerosis is a rare, progressive disease that leads to hardening and tightening of the skin and connective tissues. It usually begins with a few dry patches of skin on the hands or face that begin getting thicker and harder. These patches then spread to other areas of the skin. In some cases, systemic sclerosis also affects the blood vessels an internal organs. Systemic sclerosis is one of a group of arthritic conditions called connective tissue disorders, a person's antibodies are directed against their own tissues.

ELIGIBILITY:
Inclusion Criteria:

1. All patients must fulfill the criteria for SSc by ACR criteria
2. Age of entry into the study ≥ 18 yrs
3. FVC <85% of predicted.
4. Able to complete the 6MWT with a walking distance ≥ 150 m
5. Patients must have dyspnea on exertion (grade ≥ 2 on the Magnitude of Task component of the Mahler Modified Dyspnea Index).
6. SSc for ≤ 10 years, with onset defined as the date of the first non-Raynaud manifestation typical of systemic sclerosis.
7. Patients may have limited (cutaneous thickening distal but not proximal to elbows and knees, with or without facial involvement) or diffuse (cutaneous thickening proximal to elbows and knees, often involving the chest or abdomen) cutaneous SSc (Medsger 1995).
8. Patients must show some evidence of alveolitis as defined by an HRCT of the lung which shows ground glass opacification as a radiographic marker of "alveolitis" or finely reticulated fibrosis or they must have alveolitis by BAL ( ≥ 3% PMN's or ≥ 2% eosinophils).
9. Female patients of childbearing potential must have negative pregnancy test within 7 days before initiation of study drug dosing.
10. Patients must be able to provide written voluntary informed consent.

Exclusion Criteria:

1. FVC ≤ 50% of predicted or DLCO (corrected for Hgb but not for alveolar volume) ≤ 35% of predicted (suggesting severe probably irreparable disease and/or significant pulmonary vascular involvement by SSc).
2. FEV1/FVC ratio <65% (to exclude significant airflow obstruction)
3. Clinically significant abnormalities on HRCT not attributable to SSc (e.g., lung mass, extensive scarring due to previous infection, etc.)
4. Clinically significant pulmonary hypertension documented on right heart catheterization (i.e., right ventricular systolic pressure of >50 mm Hg and/or mean PAP ≥30 mm Hg) pulmonary pressure or echocardiographic evidence of PAH (if echo cardiographic systolic pressure ≥ 55 mmHg) or FVC/DLCO ratio >1.6 on pulmonary function testing
5. Persistent unexplained hematuria (>10 RBCs/hpf).
6. History of persistent leukopenia (white blood cell count <3500), neutropenia (absolute neutrophil count < 1500) or thrombocytopenia (platelet count <100,000).
7. Clinically significant anemia (<9.0 gm/dl)
8. Serum creatinine >ULN.
9. Pregnancy (documented by urine pregnancy test), breast feeding
10. If of child-bearing potential, failure regularly to employ a reliable means of contraception
11. Active infection of the lung or elsewhere, whose management would be compromised by Imatinib
12. Unreliability, drug abuse (including active alcoholism)
13. Any chronic, debilitating illness (other than SSc)
14. Smoking of cigars, pipes or cigarettes during the past 6 months
15. Baseline liver function tests (ALT or AST or bilirubin >1.5 x upper limit of normal
16. Previous use of prednisone > 10 mg per day. If on prednisone ≤10 mg/d, dose must have been stable for > 1 month.
17. All other medication with putative disease-modifying properties (e.g., D-penicillamine, cyclophosphamide, azathioprine, methotrexate, colchicine, Potaba) must be discontinued 1 month prior to beginning study medication.
18. Patient is < 5 years since she/he had a primary malignancy except: if the other primary malignancy is not currently clinically significant nor requiring active intervention, or if other primary malignancy is a basal cell skin cancer or a cervical carcinoma in situ. Existence of any other malignant disease is not allowed except after consultation with the PI.
19. Patient with Grade III/IV cardiac problems as defined by the New York Heart Association Criteria. (i.e., congestive heart failure, myocardial infarction within 6 months of study)
20. Patient has a severe and/or uncontrolled medical disease (i.e., uncontrolled diabetes, chronic renal disease, or active uncontrolled infection).
21. Patient has known chronic liver disease (i.e., chronic active hepatitis and cirrhosis).
22. Patient has a known diagnosis of human immunodeficiency virus (HIV) infection.
23. Use of contraindicated medications at baseline.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2007-08; Primary Completion 2008-11 (Actual); Study Completion 2008-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Daniel E. Furst, MD, Principal Investigator — University of California, Los Angeles
Locations (1):
- UCLA David Geffen School of Medicine, Division of Rheumatology, Los Angeles, California, United States

REFERENCES:
- [Result] Khanna D, Saggar R, Mayes MD, Abtin F, Clements PJ, Maranian P, Assassi S, Saggar R, Singh RR, Furst DE. A one-year, phase I/IIa, open-label pilot trial of imatinib mesylate in the treatment of systemic sclerosis-associated active interstitial lung disease. Arthritis Rheum. 2011 Nov;63(11):3540-6. doi: 10.1002/art.30548. PMID 21769849

RESULTS

PARTICIPANT FLOW:
Recruitment Details: University setting convenience samples.
Pre-assignment Details: 1-year, Phase I/IIa, Open-label trial
Groups:
- Imatinib: Systemic Sclerosis patients administered oral 600 mg imatinib once per day for up to one year.
Period: Overall Study
Arm/Group | Imatinib
Started | 20
Completed | 12
Not Completed | 8
Not completed — Adverse Event | 7
Not completed — Lost to Follow-up | 1

BASELINE CHARACTERISTICS:
Arm/Group | Imatinib
Number analyzed (Participants) | 20
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 20
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 46.1 (14.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13
  Male | 7
Region of Enrollment [Number; unit: participants]
  United States | 20

OUTCOME MEASURES:

1. Primary Outcome: Treatment-related Adverse Events
Description: Treatment-related adverse events requiring discontinuation.
Time Frame: Baseline vs. Endpoint (1 year)
Measure: Number; unit: participants
Arm/Group | Imatinib
Number analyzed (Participants) | 20
participants | 5

2. Secondary Outcome: Change in FVC (Forced Vital Capacity)
Description: Measures the amount of air breathed out as a percent of predicted.
Time Frame: Baseline vs. Endpoint (1 year)
Measure: Mean (Standard Deviation); unit: Percent predicted
Arm/Group | Imatinib
Number analyzed (Participants) | 20
Percent predicted | 1.74 (2.1)

3. Secondary Outcome: Change in TLC (Total Lung Capacity)
Description: No measures of dispersion was available for TLC as data were lost. This describes the total lung capacity as a percent of predicted.
Time Frame: Baseline vs. Endpoint (1 year)
Measure: Mean (Standard Deviation); unit: Percent predicted
Arm/Group | Imatinib
Number analyzed (Participants) | 20
Percent predicted | 4.17 (NA) — Data was lost.

4. Secondary Outcome: Change in DLco
Description: DLCO (diffusing capacity or transfer factor of the lung for carbon monoxide (CO)) is the extent to which oxygen passes from the air sacs of the lungs into the blood. Commonly, it refers to the test used to determine this parameter.
Time Frame: Baseline vs. Endpoint (1 year)
Measure: Mean (Standard Deviation); unit: Percent predicted
Arm/Group | Imatinib
Number analyzed (Participants) | 20
Percent predicted | 1.46 (NA) — Data was lost.

5. Secondary Outcome: Change in Modified Rodnan Skin Score (MRSS)
Description: No measures of dispersion was available as data were lost. The range of this measure is 0 to 51 and measures the extent of skin thickening with higher numbers representing thickening.
Time Frame: Baseline vs. Endpoint
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Imatinib
Number analyzed (Participants) | 20
units on a scale | 3.9 (NA) — Data was lost.

ADVERSE EVENTS:
Arm/Group | Imatinib
Serious Adverse Events (participants affected / at risk) | 3/20
Other Adverse Events (participants affected / at risk) | 10/20
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Imatinib (N=20)
Anemia (Blood and lymphatic system disorders) | 1 (1)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Generalized Edema (General disorders) | 2 (2)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Imatinib (N=20)
Fatigue (General disorders) | 7 (7)
Facial/lower extremity edema (Renal and urinary disorders) | 9 (16)
Nausea/Vomiting (Gastrointestinal disorders) | 9 (9)
Generalized rash (Skin and subcutaneous tissue disorders) | 4 (4)
Upper respiratory tract infection (Respiratory, thoracic and mediastinal disorders) | 4 (4)
Elevated CPK (Musculoskeletal and connective tissue disorders) | 1 (1)
Mild hemoptysis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Hypothyroidism (Endocrine disorders) | 1 (1)

LIMITATIONS AND CAVEATS:
Open label, small.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No